CLINICAL TRIAL: NCT01576965
Title: Mechanical Bowel Preparation Before Laparoscopic Hysterectomy and and Laparoscopic Sacrocolpopexy: a Randomized Controlled Trial
Brief Title: Mechanical Bowel Preparation Before Laparoscopic Hysterectomy and Laparoscopic Sacrocolpopexy: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11-1602
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2015-02

CONDITIONS: Laparoscopic Hysterectomy and/or Laparoscopic Sacrocolpopexy
Keywords: Laparoscopic hysterectomy,laparoscopic sacrocolpopexy,bowel prep
MeSH Terms: interventions — sodium phosphate

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Bowel Prep Group (Experimental): Half of the subjects will be randomized to a group that does mechanical bowel preparation with sodium phosphate enema. Those assigned to the mechanical bowel prep group will be asked to administer a single sodium phosphate enema rectally before going to bed the night before surgery. If stool is not clear in the morning, mechanical bowel prep subjects will administer one additional enema the morning of surgery. All subjects will be instructed to restrict their diet to clear liquids the day prior to their surgery and to continue this diet after midnight, save a small sip of water for medications in the morning.
  Interventions: Drug: Fleet Enema (sodium biphosphate and sodium phosphate)
- No Bowel Prep Group (No Intervention): Participants randomly assigned to this group will not have the bowel prep treatment before the surgery. All subjects will be instructed to restrict their diet to clear liquids the day prior to their surgery and to continue this diet after midnight, save a small sip of water for medications in the morning.

INTERVENTIONS:
Drug: Fleet Enema (sodium biphosphate and sodium phosphate) — Those assigned to the mechanical bowel prep group will be asked to administer a single sodium phosphate enema rectally before going to bed the night before surgery. If stool is not clear in the morning, mechanical bowel prep subjects will administer one additional enema the morning of surgery
  Arms: Mechanical Bowel Prep Group

SUMMARY:
The purpose of this study is to learn about bowel preparation (cleansing) before laparoscopic hysterectomy and/or sacrocolpopexy. We are most interested in the ability of the surgeon to view necessary anatomy for the surgery, which will be assessed by a questionnaire completed at the end of your operation by the surgeon. We hypothesize that bowel preparation before laparoscopic hysterectomy will result in improved ability of the surgeon to view necessary anatomy for the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing planned laparoscopic hysterectomy, with or without concomitant sacrocolpopexy, for benign indications with members of the Advanced Laparoscopy & Pelvic Pain division and the Urogynecology division at UNC.

Exclusion Criteria:

* Patients with known or suspected malignancy and those with severe endometriosis of the posterior cul-de-sac where bowel resection
* Pregnant women.
* Women under 18 years old.
* Women who cannot provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Surgeon's assessment of surgical field visual quality | immediately after surgery

SECONDARY OUTCOMES:
Surgeon evaluation of patient outcomes | immediately after surgery
  Survey will include questions regarding operative time, operative complications, postoperative complications, and length of hospitalization.
Patient reported satisfaction | immediately prior to surgery
  Participants will complete questionnaires regarding their relative comfort in the preoperative period. Participants will also be asked if they were able to complete the regimen and if they would be willing to perform the same preparation before a future surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Siedhoff, MD, MSCR, Principal Investigator — UNC OB-GYN Division of Advanced Laparoscopy and Pelvic Pain
Locations (1):
- UNC Department of Obstetrics and Gynecology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Siedhoff MT, Clark LH, Hobbs KA, Findley AD, Moulder JK, Garrett JM. Mechanical bowel preparation before laparoscopic hysterectomy: a randomized controlled trial. Obstet Gynecol. 2014 Mar;123(3):562-567. doi: 10.1097/AOG.0000000000000121. PMID 24499763